CLINICAL TRIAL: NCT03627676
Title: Efficacy of Cryoablation of Abdominal Wall Endometriosis: a Phase II Trial
Brief Title: Efficacy of Cryoablation of Abdominal Wall Endometriosis
Acronym: CRYOENDOMET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P160802J; 2017-A02409-44 (Other: ANSM)
Record Dates: First submitted 2018-05-29; First posted 2018-08-13 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-02

CONDITIONS: Nodule; Endometriosis
Keywords: Nodules of endometriosis; Cryoablation
MeSH Terms: conditions — Endometriosis | interventions — Cryosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental)
  Interventions: Procedure: Cryoablation

INTERVENTIONS:
Procedure: Cryoablation — Two percutaneous cryoprobes would be used for all patients. The 17-Gauge cryoprobes is introduced into the masses under US guidance. Mean distance to the skin has to be 5mm at least. Although US guidance is used, a non-enhanced CT scan may be used to assess the position of the cryoprobes before ablation, and to obtain a baseline examination in order to avoid thermal injuries to adjacent tissues such as the bowel during the ice growth. No ice extension to the skin has to be observed during cycles assessed by real-time US monitoring. Each cryoablation procedure involves 3 successive cycles: 10 minutes freeze with Argon gas, followed by 9 minutes passive and 1 minute active thawing with Helium gas, followed by a second 7 minutes freeze. The ice covered the entire targeted lesion on the short axes is visualize by US or CT-scan performed at the end of the three cycles or after repositioning. At the end of the cryoablation procedures, the probes are removed through active thawing.

SUMMARY:
The aim of this study is to evaluate for the first time prospectively the efficacy on the symptoms and the tolerance of percutaneous cryoablation performed under radiological guidance of endometriosis of the abdominal wall in alternative to surgery after validation in multidisciplinary meeting.

DETAILED DESCRIPTION:
Design of the study :

Non-comparative, non-randomized monocentric phase II trial designed as a two-staged Simon minimax plan.

Inclusions will be suspended at the end of the first stage. Statistical stopping rules are detailed in the justification of the number of patients required.

Inclusion: Patients will be included after validation in multidisciplinary consultation by the interventional radiologist in charge of the patient.

Follow-up: Only the cryoablation procedure is performed as an alternative to surgery, the usual follow-up of these patients will be maintained (1 consultation / 3 months, 1 MRI every 6 months). Additional consultations on D7 and M1 will be conducted by phone (symptoms and pain history only).

Device(s) under investigation The Endocare® Cryocare® Systems consist of a compact, easy-to-operate console and associated accessories that include Endocare® cryoprobes to deliver cold temperatures to the therapeutic tissue and Endocare® TempProbe® devices to monitor temperatures in the surrounding tissue. The Cryocare® Systems are intended for use in open, minimally invasive procedures in the areas in general surgery, urology, gynecology, oncology, neurology, dermatology, proctology, pulmonary surgery and thoracic surgery.

The systems are designed to freeze/ablate tissue by the application of extreme cold temperatures including prostate and kidney tissue, liver metastases, tumors, skin lesions, and warts.

CE Mark; Classe IIa

Expected benefits for the participants and for society This study has a direct individual benefit because of the proposed curative treatment by cryoablation as an alternative to other therapeutic modalities. For the society, the minimally invasive cryoablation may reduce the hospitalization stay and the complication's rate compare to the reference standard (surgery).

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥18 years,
* Initial radiological diagnosis of endometriosis of the abdominal wall, radiologically proven by MRI (or Doppler-ultrasound or CT-scan) with or without contrast injection,
* Symptomatic nodule (pain),
* Patient in at least one of the following situations:

  * Failure of previous treatments: recurrence of symptoms (pain) after medical therapies following the Haute Autorité de Santé (HAS) recommendations and / or prior surgery,
  * Or first-line or second-line medical therapies following the HAS recommendations considered as potentially non effective locally in multidisciplinary consultation meeting, or contraindicated or refused by patient,
  * Or surgery considered as potentially non effective locally or as a potential cause of adverse effects and morbidity because too devastating, in multidisciplinary consultation meeting,
* Cryoablation technically feasible after discussion in multidisciplinary consultation meeting:

  * localization at a distance of 5 mm from the skin (risk of skin lesion if the ice ball is at less than 5 mm from the skin) and from major nervous structures (risk of sideration),
  * 3 nodules maximum
  * nodule size up to 5 cm (<5 cm) in the largest diameter
* Absence of contraindications to general anesthesia if applicable,
* Effective contraception during participation in the study.
* Informed consent signed,
* Patient affiliated to a social security.

Exclusion Criteria:

* Pregnant woman,
* Uncontrolled coagulation disorders (TP <50%, TCA> 1.5x control) or anticoagulant therapy (blood sample prescribed at the inclusion and results verified at D0),
* Abnormalities of the hemogram: platelets <90000/mm3 (blood sample prescribed at the inclusion and results verified at D0),
* Documented infectious disease,
* Patient included in another interventional study,
* Impossibility to submit to the medical follow-up for geographical, social or psychological reasons,
* Patients deprived of liberty or subject to a legal protection measure or unable to express their consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2018-02-08 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
To evaluate the clinical efficacy at 6 months of cryoablation on the pain initially presented by the patients, pain being the principal reason of consultation. | 6 months
  The post-therapeutic pain is quantified by Numerical Scale (NS) at 6 months of cryoablation.
  Clinical success is defined as a complete response (NS= 0) or a reduction of at least 50% in the NS score at baseline.

SECONDARY OUTCOMES:
Complications rate at 6 months of cryoablation | 6 months
  The occurrence of all complications of cryoablation between the intervention and the end of follow-up, according to the classification of the NCI-CTCAE toxicity scale, will be considered.
The rate of full hospitalization after cryoablation when an outpatient basis was planned | 6 months
  Proportion of hospitalisation in woman with outpatient stay initialy planned.
The length of hospitalization (number of days) when a full hospitalization was planned | 6 months
  Total duration of hospitalization according to the type of initial stay (outpatient or hospitalization) planned, defined as the time (number of days) from the date of entry and the date of departure of the initial intervention + delays (in days) between entry date for a new intervention and date of exit within the limit of 6 Months of follow-up.
The evolution of pain (1) | baseline
  The evolution of the pain assessed at inclusion (D-90-D-3 = inclusion) by a Numerical scale.
The evolution of pain (2) | hour 0
  The evolution of the pain assessed immediately before (H0) cryoablation by a Numerical scale.
The evolution of pain (3) | 6 hours post-intervention
  The evolution of the pain assessed after cryoablation (H6) by a Numerical scale.
The evolution of pain (4) | 7 days post-intervention
  The evolution of the pain assessed at D7 by a Numerical scale.
The evolution of pain (5) | 1 month post-intervention
  The evolution of the pain assessed at 1 month by a Numerical scale.
The evolution of pain (6) | 3 months post-intervention
  The evolution of the pain assessed at 3 months by a Numerical scale.
The evolution of pain (7) | 6 months post-intervention
  The evolution of the pain assessed at 6 months by a Numerical scale.
The evolution of quality of life | baseline, 3 and 6 months post-intervention
  The evolution of the quality of life by the EHP-5 self-questionnaire. The quality of life is assessed at inclusion and at 3 and 6 months of cryoablation.
The success rate of the technique of cryoablation at 6 months | 6 months
  The technical success at 6 months is defined by a reduction in volume of endometriosis nodule of at least 2/3 of the initial volume on MRI (complete or partial response on MRI according to the RECIST criteria) at 6 months of treatment. Success rate will be assessed at the level of the treated nodule.

CONTACTS AND LOCATIONS:
Overall Officials: François Cornelis, Professor, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Radiology Department, Paris, France

IPD SHARING:
Plan to Share IPD: No